CLINICAL TRIAL: NCT03436524
Title: Development of a Prognostic Tool for Predicting Prognosis in Early Stage Chronic Lymphocytic Leukemia Patients
Brief Title: A Prognostic Tool for Early Stage CLL
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Davide Rossi, MD, PhD, Principal investigator, Oncology Institute of Southern Switzerland
Other Study IDs: IOSI-EMA-005
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Early stage CLL; Binet A; Prognosis
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Cohort of chronic lymphocytic leukemia patients at Binet A stage for the development of the risk stratification model
- Validation cohorts: Cohorts of chronic lymphocytic leukemia patients at Binet A stage for the validation of the risk stratification model

SUMMARY:
The study aims at developing a model for the prediction of time to first treatment in chronic lymphocytic leukemia patients presenting with asymptomatic early stage disease

DETAILED DESCRIPTION:
Already existing and coded health-related personal data will be retrospectively collected from the CLL databases of the Institute of Oncology Research and of the Division of Hematology of the University of Eastern Piedmont.

The adjusted association between exposure variables and time to first treatment will be estimated by Cox regression. This approach will provide the covariates independently associated with progression free survival that will be utilized in the development of a model to predict time to first treatment.

Model performance (c-index and net reclassification improvement) in discriminating patients who will eventually be treated vs patients who will not be eventually treated will be compared with that of already existing prognostic model that have been validated to predict overall survival but not time to first treatment in CLL (i.e. CLL-IPI, MDACC score, Barcelona-Brno score).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years or older
* Diagnosis of chronic lymphocytic leukemia
* Binet A stage at presentation
* No treatment need at presentation
* Availability of the baseline and follow-up annotations

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with asymptomatic chronic lymphocytic leukemia at stage Binet A.
Sampling Method: Probability Sample
Enrollment: 4933 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Discrimination capacity of the study model (per c-index) | Time to first treatment: interval between diagnosis and first line therapy (event), death without treatment (censoring), or last follow up without treatment (censoring), up to 20 years
  Primary endpoint of the study model ability in discriminating patients who will be eventually treated vs patients who will not be eventually treated.
  The discrimination capacity of the model will be assessed by calculating the c-index. This approach will allow to estimate the model accuracy and its capacity of discriminating outcome at the individual patient level. Model performance (net reclassification improvement) in discriminating patients who will be eventually treated vs patients who will not be eventually treated will be compared with that of already existing prognostic models that have been validated to predict overall survival but not time to first treatment in CLL (i.e. CLL-IPI, MDACC score, Barcelona-Brno score).

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, PhD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (1):
- Azienda Ospedaliera Universitaria Maggiore della Carità, Novara, Italy

REFERENCES:
- [Result] Condoluci A, Terzi di Bergamo L, Langerbeins P, Hoechstetter MA, Herling CD, De Paoli L, Delgado J, Rabe KG, Gentile M, Doubek M, Mauro FR, Chiodin G, Mattsson M, Bahlo J, Cutrona G, Kotaskova J, Deambrogi C, Smedby KE, Spina V, Bruscaggin A, Wu W, Moia R, Bianchi E, Gerber B, Zucca E, Gillessen S, Ghielmini M, Cavalli F, Stussi G, Hess MA, Baumann TS, Neri A, Ferrarini M, Rosenquist R, Forconi F, Foa R, Pospisilova S, Morabito F, Stilgenbauer S, Dohner H, Parikh SA, Wierda WG, Montserrat E, Gaidano G, Hallek M, Rossi D. International prognostic score for asymptomatic early-stage chronic lymphocytic leukemia. Blood. 2020 May 21;135(21):1859-1869. doi: 10.1182/blood.2019003453. PMID 32267500